CLINICAL TRIAL: NCT05049057
Title: Treatment of Acute Post-Traumatic Headache With Erenumab 140 mg, Military Service Members and Civilians With Mild TBI: A Randomized, Double Blind, Placebo Controlled, Multicenter 12-week Duration Study Followed by a 4-week Open-Label Safety Extension
Brief Title: Treatment of Acute PTH With a CGRP Receptor mAb in Military Service Members and Civilians With mTBI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNRM-CGRP-2020
Record Dates: First submitted 2021-07-26; First posted 2021-09-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Posttraumatic Headache; Mild Traumatic Brain Injury
MeSH Terms: conditions — Post-Traumatic Headache; Brain Concussion | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Drug (Experimental): Erenumab administered once monthly via two 70-mg subcutaneous injections at 3 time points over a 12-week period.
  Interventions: Drug: Erenumab 140 Mg/mL Subcutaneous Solution
- Placebo (Placebo Comparator): Placebo administered once monthly via two subcutaneous injections at 3 time points over a 12-week period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erenumab 140 Mg/mL Subcutaneous Solution — Active erenumab delivered via subcutaneous injection.
  Other Names: Aimovig
  Arms: Active Drug
Drug: Placebo — Placebo delivered via subcutaneous injection.
  Arms: Placebo

SUMMARY:
This study aims to assess the effect and safety of erenumab compared to placebo for the treatment of acute posttraumatic headache (PTH) in military service members and civilians with mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
Headache is recognized as one of the most common and disabling symptoms following head trauma. This study is designed to assess a calcitonin gene-related peptide (cGRP) monoclonal antibody (erenumab) for the preventive treatment of PTH based on the rationale that headache posttrauma is similar to migraine and is mediated by the activation of the trigeminal vascular system and subsequent release of cGRP. This study is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability, and efficacy of erenumab 140 mg for the treatment of PTH in military service members and civilians with mTBI at military treatment facilities across the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤50 years of age
* mTBI from any cause including impact, rotational acceleration, blast, or a combination, has occurred within the prior 7 days
* PTH has occurred within the prior 7 days
* Able to provide informed consent
* Likely to stay in the same geographical area for the duration of study
* Has a personal health care provider for standard of care PTH and TBI, including education, diagnostic procedures including neuroimaging and treatment, as deemed clinically indicated by the health care provider

Exclusion Criteria:

* Sustained a moderate or severe TBI, rather than mTBI, indicated with at least 1 of the following associated with head injury:

  1. abnormal structural imaging
  2. loss of consciousness for >30 minutes
  3. alteration of consciousness/mental state for >24 hours 3. post-traumatic amnesia for >1 day
* Participants with ongoing chronic migraine or other chronic daily headache disorders at the time of injury

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 404 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2027-05-19 (Estimated)

PRIMARY OUTCOMES:
Monthly Headache Days | Week 8 to Week 12
  Effect of erenumab versus placebo on monthly headache days as measured by the daily headache diary

SECONDARY OUTCOMES:
Monthly Headache Days | Week 0 to Week 12
  Effect of erenumab versus placebo on monthly headache days as measured by the daily headache diary
Monthly Headache Days | Week 0 to Week 4
  Effect of erenumab versus placebo on monthly headache days as measured by the daily headache diary
Monthly Headache Days | Week 0 to Week 8
  Effect of erenumab versus placebo on monthly headache days as measured by the daily headache diary
Adverse Events | Week 0 to Week 12
  Number of adverse events reported in erenumab group compared to placebo
Return to Full Duty | Week 0 to Week 12
  Time to return to full activity as measured by the daily headache diary
Concomitant Medications | Week 0 to Week 12
  Monthly use of medications for acute headache treatment
Headache Days | Week 0 to Week 12
  Monthly headache days after early acute versus late acute administration of erenumab compared to placebo
HPFID Activity | Week 0 to Week 12
  Monthly impact on everyday activity scores as measured by the Headache Physical Function Impact Diary Domain 1
HPFID Physical Impairment | Week 0 to Week 12
  Monthly impact on physical impairment scores as measured by the Headache Physical Function Impact Diary Domain 2
HIT-6 | Week 0 to Week 12
  Change from baseline in headache impact scores as measured by the Headache Impact Test
PHQ-9 | Week 0 to Week 12
  Change from baseline in depressive symptoms after mTBI as measured by the self-report questionnaire, Patient Health Questionnaire-9, Total Score. Total scores range from a minimum of 0 to a maximum of 27, which are rated from minimal to severe levels of depression.
ISI | Week 0 to Week 12
  Change from baseline in insomnia scores as measured by the Insomnia Severity Index

OTHER OUTCOMES:
MSQ | Week 0 to Week 12
  Change from baseline in quality of life scores as measured by the Migraine-specific Quality of Life Questionnaire
ASC-12 | Week 0 to Week 12
  Change from baseline in frequency of allodynia symptoms as measured by the Allodynia Symptom Checklist
ANAM | Week 0 to Week 12
  Change from baseline in neuropsychological functions as assessed by the Automated Neuropsychological Assessment Metrics
Function of Time | 0-24 hours, 24-72 hours, 72-144 hours
  Effect of erenumab compared to placebo as a function of time from mTBI to first dose of erenumab as measured by the daily headache diary

CONTACTS AND LOCATIONS:
Overall Officials: David L Brody, MD, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (4):
- United States (4):
  - Womack Army Medical Center - Fort Liberty, Fort Bragg, North Carolina
  - University of Pittsburgh Concussion Research Laboratory, Pittsburgh, Pennsylvania
  - William Beaumont Army Medical Center, El Paso, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Identifier-free participant data sets will be shared with the Uniformed Services University Center for Neuroscience and Regenerative Medicine Data Repository. Identifier-free data sets may also be shared with the Federal Interagency Traumatic Brain Injury Research (FITBIR) Data Repository
Time Frame: After study completion, data sets will be de-identified and shared with the repositories. De-identified data sets will be stored in the repositories indefinitely.
Access Criteria: Access to the CNRM Data Repository will be determined b the CNRM Data Quality, Access, and Publication Committee. Investigators requesting access to the data will provide a list of investigators and collaborators who will have access to the data, documentation of Ethical Conduct of Research and Human Participants Protection Training, and documentation of Institutional Review Board Approval of the research project.
  Access to FITBIR will follow FITBIR Access Criteria.
URL: http://fitbir.nih.gov/content/access-data